CLINICAL TRIAL: NCT03041038
Title: A Multicenter Study With a Randomized, Double-Blind, Placebo-Controlled Period, Followed by an Open-Label Maintenance Dosing Period to Evaluate the Efficacy and Safety of Secukinumab in Patients With Ichthyoses
Brief Title: The Efficacy and Safety of Secukinumab in Patients With Ichthyoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457AUS05T
Record Dates: First submitted 2017-01-17; First posted 2017-02-02 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Ichthyosis; Autosomal Recessive Congenital Ichthyosis; Lamellar Ichthyosis; Congenital Ichthyosiform Erythroderma; Epidermolytic Ichthyosis; Netherton Syndrome
MeSH Terms: conditions — Ichthyosis; Ichthyosis, Lamellar; Ichthyosiform Erythroderma, Congenital; Hyperkeratosis, Epidermolytic; Netherton Syndrome | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Secukinumab (Experimental): Secukinumab 300mg (liquid formation) administered subcutaneously weekly for 5 weeks then monthly until end of trial
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Placebo (sterile saline) 2ml administered subcutaneously weekly for 5 weeks then monthly until end of trial
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — Anti IL-17A antibody
  Other Names: Cosentyx
  Arms: Secukinumab
Drug: Placebo
  Other Names: Sterile Saline
  Arms: Placebo

SUMMARY:
The ichthyoses are a group of lifelong genetic disorders which share characteristics of generalized skin thickening, scaling and underlying cutaneous inflammation. There are no therapies based on growing understanding of what causes the disease. However, there have been recent discoveries of marked elevations in expression of interleukin-17A (IL-17A) and IL-17-related cytokines in the skin of individuals with ichthyosis, which may explain the inflammation. Investigators propose that IL-17-targeting therapeutics will safely suppress the inflammation and possibly the other features of ichthyosis, improving quality of life.

DETAILED DESCRIPTION:
The ichthyoses are a group of lifelong genetic disorders which share characteristics of generalized skin thickening, scaling and underlying cutaneous inflammation. The vast majority are orphan disorders and are associated with extremely poor quality of life related to social ostracism from altered appearance, associated itchiness and discomfort, and functional limitations from the skin disease. Among the most common of these orphan disorders are autosomal recessive congenital ichthyosis (ARCI) with its phenotypic subsets of lamellar ichthyosis (ARCI-LI) and congenital ichthyosiform erythroderma (ARCI-CIE), epidermolytic ichthyosis (EI) and Netherton syndrome (NS). Therapy is time-consuming for patients or parents and is supportive, focusing on clearance of the scaling. There are no therapies based on growing understanding of what causes the disease. There have been recent discoveries of marked elevations in expression of interleukin-17A (IL-17A) and IL-17-related cytokines in the skin of individuals with ichthyosis, which may explain the inflammation. Psoriasis, another inflammatory skin disorder with redness and scaling, has now been shown to result from IL-17 pathway activation and IL-17A inhibition is the most effective therapy known to treat psoriasis. Investigators propose that IL-17-targeting therapeutics will safely suppress the inflammation and possibly the other features of ichthyosis, improving quality of life. In this long-term, open-label extension, Investigators propose to treat adults with ichthyosis and at least moderate erythema with subcutaneously administered anti-IL-17 antibody (secukinumab) and to serially assess clinical response to this therapy and its safety.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent
* Subjects are at least 18 years of age or older at the time of screening
* Female subjects must not be pregnant or breast-feeding
* Female subjects of child-bearing potential with a negative urine pregnancy test and using at least one form of contraception (abstinence allowed)
* Subjects must have a confirmed diagnosis of ARCI (divided phenotypically into ARCI-LI or ARCI-CIE), EI or NS (by genotype or willingness to be genotyped)
* Subjects must be clinically judged to be immunocompetent.
* Subjects will have no allergy to secukinumab or components of the product.
* Subjects will have normal baseline laboratory testing (CMP, CBC, HIV negative, hepatitis B, C negative, QuantiFERON®-TB gold negative)
* Subjects must have an erythema score of at least 18 on IASI and an IASI-E score of 12 (at least moderate severity of erythema) at baseline

Exclusion Criteria:

* Subjects who are unable to give informed consent or assent.
* Subjects without a confirmed diagnosis ARCI, EI, or NS.
* Subjects who have a known allergy to secukinumab.
* Female subjects who are pregnant, considering becoming pregnant, or will breastfeed.
* Subjects who have prior biologic use targeting IL-17A/IL-17 receptor A or IL-12/IL-23 or who have prior use of TNF-alpha blockers.
* Subjects who have used a systemic retinoid within one month prior to initiation.
* Subjects who have used topical retinoids or keratolytics within one week prior to initiation.
* Subjects who have used emollient on the area to be biopsied in the previous 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12; Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University Department of Dermatology; Emma Guttman-Yassky, MD, PhD, Principal Investigator — Mt. Sinai Hospital Department of Dermatology
Locations (2):
- United States (2):
  - Department of Dermatology, Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Department of Dermatology Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Derived] Lefferdink R, Rangel SM, Chima M, Ibler E, Pavel AB, Kim H, Wu B, Abu-Zayed H, Wu J, Jackson K, Singer G, Choate KA, Guttman-Yassky E, Paller AS. Secukinumab responses vary across the spectrum of congenital ichthyosis in adults. Arch Dermatol Res. 2023 Mar;315(2):305-315. doi: 10.1007/s00403-022-02325-3. Epub 2022 Feb 26. PMID 35218370

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (sterile saline) 2ml administered subcutaneously weekly for 5 weeks then monthly until end of trial
  Placebo
Period: Overall Study
Arm/Group | Secukinumab | Placebo
Started | 11 | 9
Week 16 | 10 | 8
Week 32 | 9 | 8
Completed | 5 | 7
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (11.7) | 35.5 (12.7) | 34.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Ichthyosis Subtype [Count of Participants; unit: Participants]
  CIE | 3 | 2 | 5
  EI | 2 | 2 | 4
  LI | 4 | 2 | 6
  NS | 2 | 3 | 5
Site [Count of Participants; unit: Participants]
  Mount Sinai | 4 | 2 | 6
  Northwestern | 7 | 7 | 14
Weight [Mean (Standard Deviation); unit: kilograms] | 69.9 (13.5) | 75.5 (30.4) | 72.4 (22.0)
Ichthyosis Area Severity Index (IASI) [Mean (Standard Deviation); unit: units on a scale] — The IASI score was modelled after the Eczema Area and Severity Index (EASI) and Psoriasis Area and Severity Index (PASI), commonly used in clinical trials for atopic dermatitis and psoriasis, respectively. This scale measures erythema and scaling and has a range of 0-48 (sum of a max score of 24 for erythema and 24 for scaling). A higher score means worse clinical severity.
  units on a scale | 33.7 (6.5) | 36.2 (4.7) | 34.8 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Reduction at Week 16 in the Ichthyosis Area Severity Index (IASI)
Description: Primary Efficacy Endpoint. The IASI score was modelled after the Eczema Area and Severity Index (EASI) and Psoriasis Area and Severity Index (PASI), commonly used in clinical trials for atopic dermatitis and psoriasis, respectively. This scale measures erythema and scaling and has a range of 0-48 (sum of a max score of 24 for erythema and 24 for scaling). A higher score means worse clinical severity. Mean difference IASI total score at Baseline was compared to IASI total score at Week 16.
Time Frame: 16 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 11 | 9
units on a scale | 2.4 [-7.8 to 12.7] | 4.3 [-6.5 to 15.1]

2. Primary Outcome: Total Number of Bacterial or Fungal Mucocutaneous Infections Through Week 16
Description: Primary Safety Endpoint
Time Frame: 16 weeks of secukinumab/placebo double blind followed by 32 week open label treatment
Measure: Number; unit: infections
Groups:
- Open Label: Participants transitioned to open label treatment with Secukinumab300mg monthly after week 16.
Arm/Group | Secukinumab | Placebo | Open Label
Number analyzed (Participants) | 11 | 9 | 18
infections | 5 | 5 | 10

ADVERSE EVENTS:
Time Frame: 56 weeks
Arm/Group | Secukinumab | Placebo | Open Label
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/9 | 1/18
Other Adverse Events (participants affected / at risk) | 3/11 | 2/9 | 6/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Secukinumab (N=11) | Placebo (N=9) | Open Label (N=18)
Hospitalization-pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hospitalization-GERD (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Secukinumab (N=11) | Placebo (N=9) | Open Label (N=18)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Flu-like symptoms (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Otitis externa bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT03041038/Prot_SAP_000.pdf